CLINICAL TRIAL: NCT00039754
Title: A Multicenter Dosimetry Trial to Evaluate Radiation Absorbed Dose From Holmium-166-DOTMP in Patients With Multiple Myeloma
Brief Title: A Trial of Skeletal Targeted Radiotherapy Using Holmium-166-DOTMP in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: business reasons
Sponsor: Poniard Pharmaceuticals (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 0102
Record Dates: First submitted 2002-06-07; First posted 2002-06-11 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Transplant; Skeletal Targeted Radiotherapy; Holmium
MeSH Terms: conditions — Multiple Myeloma | interventions — holmium-1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetrakis(methylenephosphonic acid)

INTERVENTIONS:
Drug: Holmium-166-DOTMP

SUMMARY:
Multiple myeloma is a disease that resides primarily in the bone and has shown to be sensitive to radiation. Administration of a radiotherapy agent that targets the bone, such as Holmium-166-DOTMP, in conjunction with melphalan and an autologous stem cell transplant, may improve the patient's chance of responding to treatment. The purpose of this study is to determine the amount of Holmium-166-DOTMP that localizes in the bone and in normal organs, and to evaluate the safety and efficacy of Holmium-166-DOTMP in the treatment of patients with multiple myeloma.

DETAILED DESCRIPTION:
The purpose of this study is to estimate the radiation absorbed dose to the bone marrow and kidneys based on whole-body gamma camera image data for comparison with that obtained using mathematical models based on whole body counting from a small gamma detection device called a thyroid probe; to obtain pharmacokinetic data following administration of 166Ho-DOTMP; and to evaluate safety and efficacy in patients who receive 25 Gy targeted therapy of 166Ho-DOTMP and 200 mg/m2 melphalan followed by autologous peripheral blood stem cell transplant (PBSCT).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03